CLINICAL TRIAL: NCT05364242
Title: Open-Label Phase 2/3 Clinical Study to Investigate Safety and Immunogenicity of a Single VLA2001 Booster Vaccination in Adult Volunteers, After Receipt of Nationally Rolled Out mRNA COVID-19 Vaccines and/or Natural SARS-CoV-2 Infection
Brief Title: VLA2001 Booster in Adult Participants After Priming With mRNA COVID-19 Vaccine and/or Natural SARS-CoV-2 Infection
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VLA2001-307
Record Dates: First submitted 2022-05-04; First posted 2022-05-06 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: SARS-CoV-2 Infection
Keywords: VLA2001; SARS-CoV-2 Infection; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — VLA2001 COVID-19 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VLA2001 (Experimental)
  Interventions: Biological: VLA2001

INTERVENTIONS:
Biological: VLA2001 — whole virus inactivated SARS-CoV-2 vaccine adjuvanted with cytosine phospho-guanine (CpG)1018 in combination with aluminium hydroxide

SUMMARY:
This is a clinical study to investigate the safety, tolerability and immunogenicity of a VLA2001 booster vaccination in participants aged 18 years and older. In total approximately 275 participants are planned to be enrolled.

DETAILED DESCRIPTION:
This is a multicentric, open-label, phase 2/3 study to investigate the safety, tolerability and immunogenicity of a VLA2001 booster vaccination standard dose in adults aged ≥18 to ≤50 years or double dose in volunteers aged >50 years.

Volunteers who are either generally healthy or are with a stable medical condition will be enrolled. In total approximately 275 participants were planned to be enrolled. It was planned to enroll approximately 25% of participants who are above 65 years into the cohorts with participants above 50 years of age.

Cohorts 1B, 1C, 1D, 2B and 2D have been fully recruited. Recruitment for Cohorts 1A, 2A, 2C, and 3, has been stopped in December 2022 due to very low recruitment rates in these cohorts.

The revised study design ensures a safety follow-up of at least 6 months after the VLA2001 vaccination for all enrolled study participants.

Immunogenicity will be assessed at Visits 1 (pre-booster, Day 1) and Visit 2 (Day 15, 14 days after the booster vaccination).

Safety will be assessed up to Visit 3a (Day 180) or up to an End of Study Visit for participants who have already had their Day 180 visit before the current study amendment.

ELIGIBILITY:
Inclusion Criteria:

ALL PARTICIPANTS:

1. Participants of either gender aged 18 years and older at screening
2. Participants must have read, understood, and signed the informed consent form (ICF)
3. Medically stable
4. Participant has a Body Mass Index (BMI) of 18.0-30.0 kg/m2
5. Must be able to attend all visits of the study and comply with all study procedures
6. Women of childbearing potential (WOCBP) must be able and willing to use at least 1 highly effective method of contraception
7. WOCBPs must have a negative pregnancy test prior to the booster vaccination.

Cohort 1:

Will receive a standard dose of VLA2001 (0.5 mL), if:

* Aged between 18 years and 50 years and
* Have received two or three doses of mRNA SARS-CoV-2 vaccines and have never experienced a natural SARS-CoV-2 infection, or
* Have received two or three doses of mRNA SARS-CoV-2 vaccines and have experienced a natural SARS-CoV-2 infection.

Cohort 2:

Will receive a double dose of VLA2001 (1.0 mL), if:

* older than 50 years and
* Have received two or three doses of mRNA SARS-CoV-2 vaccines and have never experienced a natural SARS-CoV-2 infection, or
* Have received two or three doses of mRNA SARS-CoV-2 vaccines and have experienced a natural SARS-CoV-2 infection.

Cohort 3:

Will receive a standard dose of VLA2001 (0.5 mL), if:

* Aged between 18 years and 50 years and
* Have never received any SARS-CoV-2 vaccine and
* Have experienced a natural SARS-CoV-2 infection

Will receive a double dose of VLA2001 (1.0 mL), if:

* Older than 50 years and
* Have never received any SARS-CoV-2 vaccine and
* Have experienced a natural SARS-CoV-2 infection

Exclusion Criteria:

ALL PARTICIPANTS:

1. Participant is pregnant or planning to become pregnant within 3 months after booster administration
2. History of allergy to any component of the vaccine
3. Participant had close contact to persons with confirmed SARS-CoV-2 infection within 30 days prior to screening (Visit 0)
4. Participant has participated in a clinical study involving an investigational SARS-CoV-2 vaccine or has received or plans to receive a licensed SARS-CoV-2 vaccine during the duration of the study
5. Significant infection or other acute illness, including fever > 37.8 °C within 48 hours before vaccination
6. Positive SARS-CoV-2 rapid Antigen test result during screening or Visit 1
7. Participant has a known or suspected defect of the immune system, such as participants with congenital or acquired immunodeficiency, including infection with HIV, status post organ transplantation or immuno-suppressive therapy within 4 weeks prior to the expected day of vaccination (Visit 1).
8. Participant has a history of malignancy in the past 5 years other than squamous cell or basal cell skin cancer. If there has been surgical excision or treatment more than 5 years ago that is considered to have achieved a cure, the participant may be enrolled.
9. History of drug dependency or current use of drug of abuse or alcohol abuse at screening
10. Significant blood loss (> 450 mL) or has donated 1 or more units of blood or plasma within 6 weeks prior to the expected day of first vaccination (Visit 1)
11. History of clinically significant bleeding disorder (e.g., factor deficiency, coagulopathy, or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venepuncture
12. Severe and uncontrolled ongoing autoimmune or inflammatory disease, History of Guillain-Barre syndrome or any other demyelinating condition
13. Any other significant disease, disorder or finding which in the opinion of the investigator may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study

    Prior/concomitant therapy:
14. Receipt of immunoglobulin or another blood product within the 3 months before expected day of vaccination (Visit 1) in this study or those who expect to receive immunoglobulin or another blood product during this study
15. Receipt of medications to treat or prevent COVID-19 (except licensed mRNA vaccine for participants of cohort 1 and 2)
16. Receipt of any vaccine (licensed or investigational), other than licensed influenza vaccine or for medical emergencies such as tetanus or rabies exposure, within 28 days prior to the expected day of first vaccination (Visit 1)

    Others:
17. Any member of the study team or sponsor
18. An immediate family member or household member of the study's personnel

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2023-05-22 (Actual)

PRIMARY OUTCOMES:
GMT (Geometric Mean Titer) fold-rise for neutralising antibodies against SARS-CoV-2 following a single booster dose with VLA2001 | Day 15
Frequency and severity of solicited AEs (Adverse Events) (local and systemic reactions) after the VLA2001 booster vaccination | until Day 7

SECONDARY OUTCOMES:
Immune response as determined by the GMT (Geometric Mean Titer) of SARS-CoV-2-specific neutralizing antibodies | Visit 1 (Day 1) and Visit 2 (Day 15)
Proportion of participants achieving an at least 2-, 4-, 10- or 20-fold rise over baseline in terms of neutralizing antibodies to SARS-CoV-2 S-protein neutralizing antibodies | Visit 2 (Day 15)
GMT (Geometric Mean Titer) fold-rise of IgG antibodies to the SARS-CoV-2 S-protein following a single booster dose with VLA2001 | Visit 2 (Day 15)
Immune response as determined by the GMT (Geometric Mean Titer) of IgG antibodies to the SARS-CoV-2 S-protein | Visit 1 (Day 1) and Visit 2 (Day 15)
Proportion of participants achieving an at least 2-, 4-, 10- or 20-fold rise over baseline in terms of IgG antibodies to SARS-CoV-2 S-protein antibodies | Visit 2 (Day 15)
Assessment of T-cell responses from PBMCs (Peripheral Blood Mononuclear Cell) after in vitro stimulation with SARS-CoV-2 antigens using e.g. ELISpot or intracellular cytokine staining | Visit 1 (Day 1) and Visit 2 (Day 15)
Frequency and Severity of any AE (Adverse Event) | up to 4 weeks after vaccination
Frequency and Severity of unsolicited AEs (Adverse Events) | up to 4 weeks after vaccination
Frequency and severity of any unsolicited vaccine-related AE (Adverse Event) | up to 4 weeks after vaccination
Frequency and severity of any SAE (Serious Adverse Event) | up to Day 180
Frequency and severity of any AESI (Adverse Event of Special Interest) | up to Day 180

CONTACTS AND LOCATIONS:
Overall Officials: Valneva Clinical Development, Study Chair — Valneva Austria GmbH
Locations (4):
- Netherlands (2):
  - General Practitioners Research Institute (GPRI), Groningen
  - European Clinical Research Alliance on Infectious Diseases (ECRAID), Utrecht
- New Zealand (2):
  - Middlemore Clinical Trials, Auckland, Papatoetoe
  - Optimal Clinical Trials, Auckland

IPD SHARING:
Plan to Share IPD: No